CLINICAL TRIAL: NCT06486909
Title: Shunt-dependency After Aneurysmal Subarachnoid Haemorrhage - the Role of Early Hyperglycaemia in Cerebro-spinal Fluid and Blood
Brief Title: Shunt-dependency After aSAH - Role of Early Hyperglycaemia in CSF and Blood
Acronym: HCP-Glc
Status: Recruiting | Type: Observational
Sponsor: Isabel Hostettler (Other)
Collaborators: Kantonsspital Aarau (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Isabel Hostettler, PD Dr. med. Isabel Charlotte Hostettler, PhD, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: 2022-02108
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Aneurysm, Ruptured; Hyperglycemia; Hydrocephalus
Keywords: aneurysmal subarachnoid haemorrhage; hyperglycaemia; hydrocephalus; ventriculo-peritoneal shunt; extra-ventricular drain
MeSH Terms: conditions — Aneurysm, Ruptured; Hyperglycemia; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebral spinal fluid (CSF) and blood serum samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aSAH Patients: Patients with an acute ruptured intracranial aneurysm.
  Interventions: Diagnostic Test: Cerebrospinal Fluid (CSF) Sample; Diagnostic Test: Blood Serum Sample

INTERVENTIONS:
Diagnostic Test: Cerebrospinal Fluid (CSF) Sample — Samples for glucose in CSF will be taken upon EVD/LD placement until EVD/LD removal (within the first 14 days).
Diagnostic Test: Blood Serum Sample — Samples for glucose in blood serum will be completed every day, for the first 14 days.

SUMMARY:
The goal of this study is to confirm the association of early increased glucose levels in cerebro-spinal fluid (CSF) and ventriculo-peritoneal-shunt (VPS)-dependency also evaluating the influence of blood glucose on VPS dependency in patients suffering from an aneurysmal subarachnoid haemorrhage (aSAH). The main questions we aim to answer are:

* Is there an association of glucose levels on VPS dependency in patients requiring extra-ventricular-drain (EVD) placement for aSAH?
* In addition, if there is, what is the influence the course of glucose levels has on VPS dependency?

Glucose levels in CSF and serum will be measured on admission, or in case of CSF, upon EVD placement. Glucose in CSF will then be measured every day until EVD removal together with serum glucose. Follow-up will be conducted in person after 3 and 6 months.

DETAILED DESCRIPTION:
Aneurysmal SAH is a haemorrhage into the subarachnoid space associated with high mortality and morbidity. Several factors influence morbidity and therefore outcome after aSAH with HCP being one such factor. Hydrocephalus is a well-known complication after aSAH. It is thought to occur due to arachnoid adhesions as a reaction to the blood in the subarachnoid space, leading to impaired CSF absorption. Hydrocephalus is associated with an increased risk of poor clinical outcome, cognitive disturbance, and decreased functional status[3-5]. As such, HCP is associated with a significant increase in morbidity and mortality in aSAH patients and warrants treatment, preferably early. In acute HCP, diversion of CSF is conducted via insertion of an EVD. Due to the blood in the CSF, a permanent system, such as a VPS, is not inserted in the early stages as it would get blocked due to clots. If patients cannot be weaned from the EVD due to persisting HCP a VPS, is then inserted if the CSF is not too bloody anymore. Incidence of aSAH-associated HCP is up to 67%, of which about 50% end up needing a VPS. Several risk factors (ie. increased age, female sex, rebleeding, intraventricular haemorrhage, Fisher grade, and Hunt and Hess grade) have been reported. One factor, especially interesting due to its potential target as a treatment option, is hyperglycaemia. Hyperglycaemia after aSAH is common and most likely due to humeral activation including catecholamine release altering homeostasis. Previous studies have reported an association between hyperglycaemia and VPS dependency. The pathophysiological mechanism behind this potential association remains unclear but is likely due to it adhesions caused by hyperglycaemia and therefore reduction of CSF outflow potentially through higher viscosity. Inflammation, disruption of immune function and disruption of endothelial function might also play a role by decreasing reabsorption. The aim of this study is to evaluate the association of glucose levels in CSF, as well as serum (as CSF glucose is proportional to blood glucose), at prespecified time points and its association with VPS dependency in patients requiring EVD. In this step, timing of VPS insertion is going to be conducted as per our standard. Assessment of early (without trying out repeated weaning) versus late VPS insertion will only be evaluated once the association has been proven in our study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Hospital admission due to an aneurysmal subarachnoid haemorrhage (radiological confirmation needed)

Exclusion Criteria:

* Younger than 18 years old
* Non-aneurysmal subarachnoid haemorrhage (eg. trauma, perimesencephalic subarachnoid haemorrhage, mycotic or flow-associated aneurysms)
* Previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with aneurysmal subarachnoid haemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Ventriculo-peritoneal shunt (VPS) dependency | 6 months
  Glucose levels in patients requiring EVD/LD placement for aSAH and its influence on VPS dependency.

SECONDARY OUTCOMES:
Modified Ranking Scale (mRS) | 6 months
  Modified Ranking Scale 0-6 where 0 means no symptoms and 6 death (adjusting for VPS dependency) in aSAH patients requiring EVD/LD placement

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Hostettler, MD PhD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (3):
- Switzerland (3):
  - Cantonal Hospital Aarau, Aarau
  - University Hospital Basel, Basel
  - Cantonal Hospital St Gallen, Sankt Gallen